CLINICAL TRIAL: NCT05061914
Title: Surgical Options for Management of Pericardial Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Omar Ragheb, resident at cardiothoracic surgery department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-09-04
Record Dates: First submitted 2021-09-20; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Pericardial Effusion
MeSH Terms: conditions — Pericardial Effusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- pericardiocentesis (Active Comparator): vitally unstable patients with tamponading pericardial effusion undergone percutaneous gradual drainage by a central venous catheter
  Interventions: Procedure: pericardial effusion drainage
- subxiphoiodal drainage (Active Comparator): drainage of the pericardial effusion through a subxiphoidal midline incision
  Interventions: Procedure: pericardial effusion drainage
- thoracotomy (Active Comparator): encysted and undiagnosed pericardial effusion drainage through anterior thoracotomy performing a pericardiopleural window and take a pericardial biopsy
  Interventions: Procedure: pericardial effusion drainage
- VATS drainage (Active Comparator): encysted and undiagnosed pericardial effusion drainage through VATS that permits performing a pericardiopleural window and take a pericardial biopsy with minimal incisions
  Interventions: Procedure: pericardial effusion drainage

INTERVENTIONS:
Procedure: pericardial effusion drainage — tamponading pericardial effusion is a life threatenning condition , pericardiocentesis is performed for patients who are vitally unstable and with a massive amount of effusion to prevent cardiac tamponade, Surgical drainage of pericardial effusion was classically conducted by either open thoracotomy or subxiphoid pericardiectomy. Thoracoscopy has established itself as an alternative to open thoracotomy for the management of many pericardial, pleural and pulmonary disorders

SUMMARY:
This is a retrospective descriptive study which will be conducted at Sohag university Hospital, Sohag, Egypt at emergency and cardiothoracic department . It includes all patients with pericardial effusion who diagnosed as temponading pericardial effusion or threatened cardiac temponade , The aim of this work is to clarify the suitability and individualization of each surgical procedure (either subxiphoidal drainage, drainage through thoracotomy or video-assisted thoracoscopic (VATS) pericardiotomy) in treatment and diagnosis of patients presenting with pericardial effusion .

DETAILED DESCRIPTION:
The normal pericardial space contains up to 50 ml of fluid that formed of a plasma ultrafiltrate and the amount greater than this amount is considered as a pathologic effusion.

The curvilinear pressure-volume relationship of the pericardial sac leads to the consequences of the pericardial effusion specially the rapidly accumulating fluid that causes cardiac tamponade.

There is a lot of diseases and complications that vary in causing pericardial effusion e.g idiopathatic pericarditis, malignancy, connective tissue diseases and heamorrhage. The management of pericardial effusion depends on whether there is tamponade or not.

Despite the new diagnostic strategies and the recent data have improved our ability to assess the presence and the amount of pericardial effusion, and assess the cause and its heamodynamic impact, the optimal management of the pericardial effusion is still controversial. While the Echocardiography is the corner stone in the management, multimodal imaging strategies specially computed tomography are dependable. The optimal therapy for symptomatic pericardial effusions remains controversial. In general, there are surgical based approaches and percutaneous-based approaches to pericardial fluid drainage.

A surgical subxiphoid approach for draining a pericardial effusion was first described in 1829 and there have been several additional methods proposed for surgical pericardial effusion drainage since that time.

In 1986, Kopecky and colleagues reported the first percutaneous pericardiocentesis series with multiple subsequent reports characterizing the relative safety and efficacy of a percutaneous approach.

Initially, pericardial effusion is classified by the volume of effusion. The treatment is directed at the primary disease in patients with a small amount of effusion without symptoms. In contrast, pericardiocentesis is performed for patients who are vitally unstable and with a massive amount of effusion to prevent cardiac tamponade, Surgical drainage of pericardial effusion was classically conducted by either open thoracotomy or subxiphoid pericardiectomy.

Thoracoscopy has established itself as an alternative to open thoracotomy for the management of many pericardial, pleural and pulmonary disorders. Thoracoscopic cardiac procedures have been performed less frequently. It affords excellent visualization of the pericardial surface, thus allowing the safe performance of pericardial resection and formation of a pericardial window.

A pericardial window allows drainage of pericardial fluid into the adjacent space, usually the pleural cavity. The subxiphoid approach is erroneously referred to as a "window" because no connection is made to the adjacent space during the standard subxiphoid approach.

The thoracoscopic approach creates a true window but it is done under general anaesthesia with single-lung ventilation and through 2 or 3 intercostal ports. However, the role of the thoracoscopic approach is limited in patients with hemodynamically significant pericardial effusions due to the positioning of the patients in the lateral decubitus which makes emergency pericardiocentesis very difficult.

Recently , video-assisted thoracoscopic (VATS) pericardiotomy has gained popularity as a minimally invasive approach. VATS allows for visual evaluation of the pericardium and is used when the diagnosis of pericardial effusion has remained undiagnosed despite previous, less-invasive tests. It is also used to drain the excess fluid and prevent its reaccumulation.

Choosing the best surgical approach to drain the pericardial effusion is a matter of debate and it should be based upon the effectiveness of the approach in avoiding recurrence of the pericardial effusion and upon the morbidity and mortality associated with the procedure. Moreover, the relative simplicity of the procedure and its cost are other important aspects that should be considered when choosing the optimal surgical approach.

ELIGIBILITY:
Inclusion Criteria:

Suspected malignant effusion . Systemic collagen diseases e.g; SLE , Rheumatoid Artheritis …… Suspected cases of tuberculosis .

Exclusion Criteria:

Cardiac tamponade as a complication of acute coronary syndromes Cardiac tamponade as a complication of aortic dissection . Pericardial effusion following penetrating and blunt chest trauma (heamopericardium).

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
recurrence | 3 months
  if there is a recurrence or not

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

REFERENCES:
- [Background] Chiabrando JG, Bonaventura A, Vecchie A, Wohlford GF, Mauro AG, Jordan JH, Grizzard JD, Montecucco F, Berrocal DH, Brucato A, Imazio M, Abbate A. Management of Acute and Recurrent Pericarditis: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jan 7;75(1):76-92. doi: 10.1016/j.jacc.2019.11.021. PMID 31918837
- [Background] Saltzman AJ, Paz YE, Rene AG, Green P, Hassanin A, Argenziano MG, Rabbani L, Dangas G. Comparison of surgical pericardial drainage with percutaneous catheter drainage for pericardial effusion. J Invasive Cardiol. 2012 Nov;24(11):590-3. PMID 23117314
- [Background] Azarbal A, LeWinter MM. Pericardial Effusion. Cardiol Clin. 2017 Nov;35(4):515-524. doi: 10.1016/j.ccl.2017.07.005. PMID 29025543